CLINICAL TRIAL: NCT01072591
Title: A Phase I, Double-blind, Randomised, Placebo-controlled, Parallel-group Study to Assess Safety,Tolerability, Pharmacokinetics and Efficacy of MEDI-578, an Anti-NGF Monoclonal Antibody, After Single Ascending Doses in Male and Non-fertile Female Patients With Painful Osteoarthritis of the Knee
Brief Title: Study to Assess MEDI -578 in Patients With Osteoarthritis (OA) of the Knee
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Amended clinical development plan.
Sponsor: AstraZeneca (Industry)
Collaborators: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D2460C00001
Record Dates: First submitted 2010-02-19; First posted 2010-02-22 (Estimated); Last update posted 2013-01-29 (Estimated); Status verified 2013-01

CONDITIONS: Osteoarthritis; Pain
Keywords: anti-NGF; OA; pain
MeSH Terms: conditions — Osteoarthritis; Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: MEDI-578
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo for MEDI-578

INTERVENTIONS:
Drug: MEDI-578 — intravenous infusion, once
  Arms: 1
Drug: Placebo for MEDI-578 — Intravenous infusion, once
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of a single intravenous dose of MEDI-578, a monoclonal antibody, in patients with osteoarthritis of the knee. It will also be evaluated how MEDI-578 is absorbed and distributed through the body.

ELIGIBILITY:
Inclusion Criteria:

* Patients with painful osteoarthritis of the knee.
* The pain from the knee must exceed pain experienced from any other condition.
* Patients must be willing and able to discontinue all current analgesic treatment.

Exclusion Criteria:

* Any other form of arthritis than osteoarthritis.
* Presence of neuropathic pain, or fibromyalgia, or wide spread chronic pain not related to osteoarthritis.
* Significant abnormalities on the clinical examination that may interfere with the study or present a safety risk to the patient, as judged by the investigator.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2010-02; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Safety variables (adverse events, vital signs, ECG, safety lab) | Assessments performed at (predose then ranging from 15 minutes to every 12 hours) on Days -1 to Day 2. Thereafter weekly assessments until week 4 when a fortnightly schedule is followed until week 8. A final assessment at week 12.

SECONDARY OUTCOMES:
To characterize the pharmacokinetics of MEDI-578 in plasma. | Blood sampling performed at (predose, then ranging from every hour to every 24 hour) on Day 1 and 2. Thereafter weekly blood sampling until week 4, when a fortnightly schedule is followed until week 8. A final assessment at week 12.
To assess the immunogenicity of MEDI-578 | Blood samples taken fortnightly from Day 1 until week 12.
To evaluate the analgesic efficacy of MEDI-578 during the night and day. | Patients will record their pain intensity every morning and evening during the 13 weeks study period.

CONTACTS AND LOCATIONS:
Overall Officials: Rolf Karlsten, Study Director — AstraZeneca RD Södertälje
Locations (1):
- Research Site, London Bridge, Greater London, United Kingdom